CLINICAL TRIAL: NCT02728232
Title: Internal Iliac Artery Ligation and Abnormally Invasive Placenta
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Mahmoud Hussein, Lecturer of Obstetrics and Gynecology, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PP2302019
Record Dates: First submitted 2016-03-31; First posted 2016-04-05 (Estimated); Last update posted 2017-04-18 (Actual); Status verified 2017-04

CONDITIONS: Placenta Percreta
MeSH Terms: conditions — Placenta Accreta

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Internal Iliac artery ligation group (Experimental): in this group the patients will undergo bilateral internal iliac artery ligation prior to the hysterectomy procedure
  Interventions: Procedure: internal iliac artery ligation; Procedure: Cesarean Hysterectomy
- Hysterectomy only (Active Comparator): in this group patients will undergo cesarean hysterectomy only
  Interventions: Procedure: Cesarean Hysterectomy

INTERVENTIONS:
Procedure: internal iliac artery ligation
  Arms: Internal Iliac artery ligation group
Procedure: Cesarean Hysterectomy

SUMMARY:
This trial is set to detect the impact of bilateral internal iliac artery ligation on the amount of intra-operative blood loss during the hysterectomy procedure done for the management of abnormally invasive placenta

ELIGIBILITY:
Inclusion Criteria:

* females with pre-operative diagnosis of abnormally invasive placenta

Exclusion Criteria:

* refusal to get enrolled in the study

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2017-04-01 (Actual); Study Completion 2017-04-01 (Actual)

PRIMARY OUTCOMES:
amount of intra-operative hemorrhage | 2-3 hours

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed M Hussein, MD, Principal Investigator — Cairo University
Locations (1):
- Kasr el aini hospital, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided